CLINICAL TRIAL: NCT02293928
Title: Impact of Hybrid Coronary Revascularization on Antiplatelet Effect of Aspirin and Clopidogrel
Brief Title: Impact of Hybrid Coronary Revascularization on Antiplatelet Therapy
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital Skejby (Other)
Collaborators: Danish Heart Foundation (Other); Aase and Ejnar Danielsens Foundation (Other)
Responsible Party: Principal Investigator, Ivy Modrau, Junior Consultant, Aarhus University Hospital Skejby
Other Study IDs: 10-000439
Record Dates: First submitted 2014-11-13; First posted 2014-11-19 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Coronary Artery Disease
Keywords: Hybrid coronary revascularization; Antiplatelet therapy; Aspirin; Clopidogrel
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 4 ml serum and 4 ml sodium citrate plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Elective hybrid coronary revascularization: All patients are treated with non-enteric coated aspirin 75 mg once daily prior to study participation. Aspirin treatment is discontinued 8-10 days prior to surgery and resumed 6-9 hours after surgery. Left internal mammary grafting of the left descendent coronary artery is performed off-pump through an inferior J-hemisternotomy (JOPCAB). All patients receive an oral loading dose of aspirin 300 mg 6-9 hours after surgery followed by daily maintenance doses of 75 mg aspirin. An oral loading dose of clopidogrel 300 mg 12 hours prior to PCI is followed by daily maintenance doses of 75 mg for 12 months. Patients are followed for 1 year.
  Interventions: Procedure: Hybrid coronary revascularization

INTERVENTIONS:
Procedure: Hybrid coronary revascularization — Hybrid coronary revascularization with standard double antiplatelet therapy

SUMMARY:
The effect of antiplatelet therapy is impaired among patients, who recently underwent on-pump coronary artery bypass grafting. The impact of hybrid coronary revascularization using minimal invasive surgical techniques on the antiplatelet effect of aspirin and clopidogrel remains unclear.

The aim of the study is to describe the impact of hybrid coronary revascularization on the effect of aspirin and clopidogrel. Furthermore, we will investigate whether high baseline platelet aggregation, high postoperative levels of platelet turnover and acute-phase response may contribute to the effect.

DETAILED DESCRIPTION:
Objective:

The effect of antiplatelet therapy is impaired among patients, who recently underwent on-pump coronary artery bypass grafting. The impact of hybrid coronary revascularization using minimal invasive surgical techniques on the antiplatelet effect of aspirin and clopidogrel remains unclear.

We hypothesize that hybrid coronary revascularization is associated with a transiently reduced antiplatelet effect of aspirin and clopidogrel. We hypothesize that the reduced antiplatelet effect of aspirin and clopidogrel could be explained by increased platelet turnover with an increased fraction of immature platelets in the peripheral blood. Furthermore, we hypothesize that the reduced antiplatelet effect is associated with increased inflammatory markers in the early postoperative phase. We hypothesize, that high platelet aggregation prior to the intervention is associated with reduced effect of antiplatelet therapy following hybrid coronary revascularization.

Methods:

40 patients with coronary artery disease will be enrolled in this prospective cohort study (recruited from a prospective pilot study conducted to assess feasibility and safety of hybrid coronary revascularization combining minimally invasive off-pump coronary artery bypass grafting through an inferior J-hemisternotomy (JOPCAB) with percutaneous coronary intervention - Clinicaltrials.gov identifier: NCT01496664). Demographics and medical history are documented preoperatively. The predicted mortality is assessed by means of the logistic European System for Cardiac Operative Risk Evaluation (EuroSCORE) I. Adverse cardiovascular events are recorded prospectively, including graft dysfunction, myocardial infarction, stroke, and pulmonary embolism.

Six blood samples are obtained from each patient:

* Pre-OP: in the outpatient setting while patients were on aspirin 75 mg daily
* Baseline: in the morning prior to surgery after eight to ten days of aspirin discontinuation (off-aspirin)
* Post-OP: on the first postoperative day when aspirin had been resumed
* Pre-PCI: on the day prior to PCI
* Post-PCI: on the first day after PCI following initiation of dual antiplatelet therapy
* 1-year follow-up: when patients were still on maintenance aspirin 75 mg and clopidogrel 75 mg Platelet function analyses are performed using Multiplate® Analyzer (Roche, Roche Diagnostics, Mannheim, Germany), VerifyNow® Aspirin, and VerifyNow® P2Y12 (Accumetrics Inc., San Diego, CA, USA). For Multiplate® Analyzer, arachidonic acid (1.0 mM) and adenosine diphosphate (6.4 and 20 uM) are used as agonists.

Complete blood counts, including immature platelet fraction (IPF), immature platelet count (IPC), and mean platelet volume (MPV), are performed using a Sysmex XE-5000 haematology analyzer (Sysmex, Kobe, Japan) with upgraded software (XE IPF Master, Sysmex) enabling flow cytometric detection of the IPF. Enzyme-linked immunosorbent assays are used according to the manufacturers' instructions to measure serum thromboxane B2 (Cayman Chemical, Ann Arbor, MI, USA) and thrombopoietin (R&D Systems Europe, Abingdon, UK). Plasma C-reactive protein was measured by immunoprecipitation using the Cobas® 6000 (Roche, Basel, Switzerland). Von Willebrand factor (antigen) and coagulation factor VIII (functional) are measured using the ACL TOP (ILS Laboratories, Bedford, MA, USA).

ELIGIBILITY:
Inclusion Criteria:

* symptomatic multivessel coronary artery disease
* treatment with non-enteric coated aspirin 75 mg once daily

Exclusion Criteria:

* aspirin or clopidogrel intolerance
* conditions prohibitive of aspirin discontinuation prior to surgery
* use of anticoagulants or any drugs other than aspirin known to affect platelet function
* use of immunosuppressive drugs
* platelet count <100 or >450 x 109/l
* inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease scheduled for elective hybrid coronary revascularization. The study cohort is recruited from a prospective pilot study conducted to assess feasibility and safety of hybrid coronary revascularization combining minimally invasive off-pump coronary artery bypass grafting and percutaneous coronary intervention (PCI) performed three to five days later (Clinicaltrials.gov identifier: NCT01496664).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Change in aspirin antiplatelet effect from preoperative to three days postoperative | 12-14 days
  Platelet aggregation measured by VerifyNow® Aspirin and Multiplate® Analyzer

SECONDARY OUTCOMES:
Change on aspirin antiplatelet effect from 3 days postoperative to 1 year follow-up | 1 year
  Platelet aggregation measured by VerifyNow® Aspirin and Multiplate® Analyzer
Change on clopidogrel antiplatelet effect from first day after PCI to 1 year follow-up | 1 year
  Platelet aggregation measured by VerifyNow®P2Y12 and Multiplate® Analyzer
Association between baseline platelet aggregation (off-aspirin) and aspirin antiplatelet effect | 12-14 days
  Platelet aggregation measured by VerifyNow® Aspirin and Multiplate® Analyzer Baseline aggregation is compared to aggragation preoperatively (on maintenance aspirin treatment) and postoperatively (when aspirin is resumed).
Correlation between acute phase reactants and platelet aggregation | 8-10 days preoperative until 1 year postoperative
  C-reactive protein, von Willebrand factor (antigen), and coagulation factor VIII (functional)
Correlation between platelet turnover and platelet aggregation | 8-10 days preoperative until 1 year postoperative
  Platelet turnover assessed by Complete blood counts, including immature platelet fraction, immature platelet count, mean platelet volume and thrombopoietin.

OTHER OUTCOMES:
Compliance to aspirin treatment at enrollment | 8-10 days preoperative
  measured by levels of serum thromboxane B2 below 30 ng/ml
Compliance to aspirin treatment at 1 year follow-up | 1 year
  measured by levels of serum thromboxane B2 below 30 ng/ml

CONTACTS AND LOCATIONS:
Overall Officials: Ivy S Modrau, MD, DMSc, Principal Investigator — Aarhus University Hospitak Skejby
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Derived] Modrau IS, Wurtz M, Kristensen SD, Hvas AM. Reduced Effect of Aspirin and Clopidogrel Following Hybrid Coronary Revascularization. Clin Appl Thromb Hemost. 2015 Oct;21(7):603-11. doi: 10.1177/1076029615573304. Epub 2015 Mar 9. PMID 25753965